CLINICAL TRIAL: NCT02953327
Title: Testing if BCG (Bacille Calmette-Guérin) Vaccination Can Induce Innate Immune Training in Adult People Above 50 Years of Age in Guinea-Bissau
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: BCGadult
Record Dates: First submitted 2016-10-21; First posted 2016-11-02 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Innate Immunity; Bacille Calmette-Guérin
Keywords: Non-Specific Effect of Vaccine; Middle aged; Immunity, heterologous

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Intervention arm, these participants will receive BCG vaccination.
  Interventions: Biological: Bacille Calmette-Guerin
- Placebo arm (Placebo Comparator): The placebo arm will receive BCG solvent.
  Interventions: Biological: BCG solvent

INTERVENTIONS:
Biological: Bacille Calmette-Guerin — Vaccine against tuberculosis
  Other Names: BCG
  Arms: Intervention arm
Biological: BCG solvent — Simple solvent
  Other Names: Diluent
  Arms: Placebo arm

SUMMARY:
The propose is to test innate immune training in a pilot study of 40 adults >50 years of age people in Guinea-Bissau. The hypothesis is that BCG vaccination will be associated with increased innate immune training measured as increased cytokine release after in vitro Peripheral Blood Mononuclear Cells (PBMC) stimulation with e.g. Mycobacterium Tuberculosis, Staphylococcus Aureus, Candida Albicans and Streptococcus Pneumoniae.

DETAILED DESCRIPTION:
BCG was developed as a vaccine against tuberculosis (TB), but many studies have now confirmed its ability to induce potent protection against other infectious diseases in children. It has recently been shown that this may be linked to increased response of the innate immune system to several non-specific pathogens after BCG exposure, so called 'innate immune training'. This training ability of BCG has been shown for children and young adults. However, to our knowledge, no studies on the ability of BCG to induce innate immune training in adults >50 years of age have been conducted. Immune training in elderly is of interest since with increasing age, the immune system gets weaker, and responds less adequately to a number of infections, for instance influenza. Thus, if BCG is able to stimulate the innate immune system in mature adults as well, it could potentially reduce the risk of serious infections in elderly.

To investigate whether BCG has innate immune training effects in mature adults, a randomized pilot study of 40 adults >50 years of age in Guinea-Bissau will be conducted. The Bandim Health Project has conducted multiple large-scale RCT's and demographic surveillance. HIV negative adults >50 years of age in a recent HIV survey are eligible for the present study. They will be checked for clinical signs of TB and an HIV test will be preformed before enrolment. Exclusion criteria are BCG vaccination within the last 10 years, illness within the last 14 days, clinical signs of active TB, and/or a positive HIV test. Those who are overtly ill will be treated or referred to hospital if needed. Those with signs of TB will be referred to the TB hospital for further examinations. Those who have become HIV positive since they were tested in the survey will receive immediate counselling and be referred to the HIV clinic.

Participants will be randomized to either BCG vaccination or placebo. To test the innate immune system blood will be withdraw 3 times: before the intervention, 2 weeks and 3 months after the intervention. There is a maximum of 10 ml blood each time, plus 3 ml the first time for the Quantiferon. This is a small volume, with a maximum of 33 ml and should not cause any problems for participants. Quantiferon results will be used as a baseline to test if participants are sensitized to mycobacterium Tuberculosis. In the blood, the innate immune training effects of BCG we will investigated by studying how the immune cells respond when they are stimulated with bacteria or other pathogens, which can cause serious infections. Provided that BCG shows induced innate immune training in adults >50 years of age, a large randomized control trial will follow to see if BCG vaccination reduces the number of acute infections in adults >50 years of age in Guinea-Bissau.

ELIGIBILITY:
Inclusion Criteria:

* adults above 50 years of age

Exclusion Criteria:

* Participants who received BCG in the last 10 years will be excluded.
* Adults who were mild to severe ill in the last 2 week will be excluded.
* Adults how have been in contact with the health system (hospital or health center) for the last 14 days will be excluded.
* People that show signs of overt disease will not be enrolled, but treated according to local standards and invited back when better.
* If the person has any sign of TB, they will excluded and be referred to the TB clinic for further investigations and treatment.
* All participants will be tested for HIV. If the test is positive, they will have an opportunity to talk with a psychologist, and we will refer them to the HIV clinic. HIV positive persons will be excluded from the present study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Change in cytokine level at 2 weeks compared to the baseline | 2 weeks
  Before intervention and 2 weeks after, blood will be withdrawn and the PBMC will be isolated. In vitro stimulation of the PBMC will be done with e.g. Mycobacterium Tuberculosis, Staphylococcus Aureus, Candida Albicans and Streptococcus Pneumoniae for 24h and 7 days. After this the cytokine levels will be measured.

SECONDARY OUTCOMES:
Change in cytokine level at 3 months compared to the baseline | 3 months
  Before intervention and 3 months after the intervention, blood will be withdrawn and the PBMC will be isolated. In vitro stimulation of the PBMC will be done with e.g. Mycobacterium Tuberculosis, Staphylococcus Aureus, Candida Albicans and Streptococcus Pneumoniae for 24h and 7 days. After this the cytokine levels will be measured. The cytokine level 3 months after intervention is the secondary outcome.

OTHER OUTCOMES:
Difference in percentage before and after BCG vaccination of a specific marker on a specific gene (e.g. H3K4me3 on TNF (tumor necrosis factor) gene). | 2 weeks and 3 months after inclusion
  Measurement of change in epigenetics after intervention, compared to before intervention.
Consultation | 3 months
  The amount of consultations in the 3 months we follow the participants. To see if there is a difference between the 2 interventions.
Medication use | 3 months
  The amount of medication use in the 3 months we follow the participants. To see if there is a difference between the 2 interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Bandim Health Project, Bissau, Bissau Codex, Guinea-Bissau

REFERENCES:
- [Derived] Berendsen MLT, Bles P, de Bree LCJ, Jensen KJ, Jensen CC, Wejse C, Mendes DV, Netea MG, Benn CS. Bacillus Calmette-Guerin vaccination induces a trained innate immunity phenotype in adults over 50 years of age: A randomized trial in Guinea-Bissau. Vaccine. 2024 Dec 2;42(26):126439. doi: 10.1016/j.vaccine.2024.126439. Epub 2024 Oct 17. PMID 39423450